CLINICAL TRIAL: NCT06449131
Title: Persistent Pleural Effusion Treatment Following Cardiothoracic Surgery by Platelet-Fibrin Glue: A Clinical Trail
Brief Title: Persistent Pleural Effusion Treatment Following Cardiothoracic Surgery by Platelet-Fibrin Glue
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daryoush Hamidi Alamdari, PhD (Other)
Responsible Party: Sponsor-Investigator, Daryoush Hamidi Alamdari, PhD, Associate professor, Mashhad University of Medical Sciences
Organization: Mashhad University of Medical Sciences (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IR.MUMS.MEDICAL.REC.981289
Record Dates: First submitted 2024-05-12; First posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Pleural Effusion
Keywords: Pleural Effusion; Persistent; Cardiac surgery; PRP; Fibrin Glue
MeSH Terms: conditions — Pleural Effusion | interventions — Fibrin Tissue Adhesive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients referred to the cardiac surgery clinic (Other): This clinical trial focused on patients referred to the cardiac surgery clinic of Imam Reza Hospital in Mashhad 2023 who were diagnosed with unilateral or bilateral pleural effusion resistant to conservative management.
  Interventions: Drug: Platelet-Rich Plasma and Fibrin Glue

INTERVENTIONS:
Drug: Platelet-Rich Plasma and Fibrin Glue — Allogenic platelet-rich plasma with fibrin glue (PRP-FG) was derived from blood obtained from a blood bank. Peripheral blood (400 ml) was collected from a donor with a matching ABO blood type, and rigorous viral safety tests were conducted. Concentrated PRP (10 ml) was obtained by subjecting the sample to centrifugation at 4000 g for 15 min to separate the plasma from the sedimented platelets.
  Fibrinogen was extracted from the separated plasma using cryoprecipitation. After freezing at -70°C followed by thawing at 4°C, fibrinogen concentrate (20 ml) was prepared by centrifugation at 6500 × g for 5 min. The concentrated PRP was combined with fibrinogen (30 ml).
  Thrombin was generated from the plasma isolated during the second centrifugation step. The ionic strength and pH were adjusted to precipitate prothrombin. The resulting precipitate was separated by centrifugation and dissolved in a calcium ion solution, resulting in a final volume of 5 ml of thrombin solution.

SUMMARY:
Persistent pleural effusion is a life-threatening complication after cardiac surgery. The traditional treatment is chest tube drainage, which may not respond to treatment. This study introduces a new noninvasive approach for treating persistent pleural effusion using platelet-rich plasma fibrin glue (PRP-FG). This method has been successfully applied for the treatment of postoperative persistent chylothorax and pneumothorax in previous studies, which significantly decreased morbidity, mortality, and hospital stay.

DETAILED DESCRIPTION:
This pilot clinical trial recruited 19 patients at Imam Reza Hospital in Mashhad, Iran (2023) who had developed unilateral or bilateral refractory postoperative effusion resistant to conventional thoracostomy treatment. Treatment success was defined as effusion <50 ml/day after 48 hours, along with symptomatic improvement and no adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of pleural effusion after cardiac surgery in open-heart surgery
* patients who sign an informed consent form

Exclusion Criteria:

* Hemodynamically unstable patients
* Patients who did not sign an informed consent form

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
The rate of air leak that is assessed by Cerfolio classification of the air leak by a single observer | within 48 hours after application of platelet-rich plasma
  Continuous: Air leak is Present throughout the respiratory cycle Inspiratory: Present during the inspiration phase of the respiratory cycle.
  Expiratory: Present only during the expiratory phase of the respiratory cycle Forced expiration: Present only when the patient coughs or forces exhalation.
Rate of radiolucency | within 48 hours after application of platelet-rich plasma
  The percent area on chest x-ray is almost completely transparent to radiation.
Patient hospitalization time | From the time the patient is admitted to the hospital to the time of discharge
  Duration of the patient's stay in hospital, assessed up to 40 weeks
Percentage of patients completely recovered | Through study completion, an average of 40 weeks
  The treatment was successful if the bubbling was stopped and lung expansion was done.
Percentage of untreated patients who died | Through study completion, an average of 40 weeks
  The bubbling was not stopped, lung expansion was not done and the patient was expired
The number of injections until the bubble stops | Through study completion, an average of 40 weeks
  PRP-FG (5-7 ml/ kg) was injected into the pleural space through the chest tube.

CONTACTS AND LOCATIONS:
Overall Officials: Daryoush Hamidi-Alamdari, Ph.D, Study Chair — Mashhad university of medical sience
Locations (1):
- Mashhad University of Medical Sciences, Mashhad, Razavi Khorasan Province, Iran

IPD SHARING:
Plan to Share IPD: No